CLINICAL TRIAL: NCT05288205
Title: A Phase 1/2a Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of JAB-21822 in Combination With JAB-3312 in Patients With Advanced Solid Tumors Harboring KRAS p.G12C Mutation
Brief Title: Phase 1/2a Study of JAB-21822 Plus JAB-3312 in Patients With Advanced Solid Tumors Harboring KRAS p.G12C Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-1006
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: KRAS P.G12C; Non-small Cell Lung Cancer; Colorectal Cancer; Pancreatic Ductal Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation (Experimental)
  Interventions: Drug: JAB-21822; Drug: JAB-3312
- Dose expansion (Experimental)
  Interventions: Drug: JAB-21822; Drug: JAB-3312

INTERVENTIONS:
Drug: JAB-21822 — KRAS G12C inhibitor
Drug: JAB-3312 — SHP2 inhibitor

SUMMARY:
This is a multicenter, open-label phase 1/2a study consisting of two parts: dose escalation phase and dose expansion phase. The objective of the dose escalation phase is to evaluate the safety, tolerability and pharmacokinetics of JAB-21822 in combination with JAB-3312 in patients with advanced solid tumors harboring KRAS p.G12C mutation and to determine the RP2D for the combination therapy. In the dose expansion phase, preliminary efficacy and safety of the combination therapy at the RP2D will be further explored in patients with specific cancer harboring KRAS p.G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent should be signed by a subject or his/her legal representative before any study-related procedures are performed;
* Subjects with histologically or cytologically confirmed locally advanced or metastatic advanced solid tumors harboring KRAS p.G12C mutation who have failed or lack standard-of-care (SOC) or are unwilling to undergo or intolerant to SOC;
* Expected survival ≥ 3 months;
* Subjects must have at least one measurable lesion as defined by RECIST v1.1. If no measurable lesion untreated with radiation is selected as the target lesion, a lesion treated with radiation ≥ 4 weeks before the first dose and with progression confirmed by radiography may be selected as the target lesion;
* Eastern Cooperative Oncology Group(ECOG) performance status 0-1;
* The organ functions of subjects meet the criteria for the following laboratory parameters at screening;
* Subjects must be able to swallow oral medications without gastrointestinal abnormalities that significantly affect drug absorption

Exclusion Criteria:

* Patients with previous (≤ 3 years) or current tumors of other pathological types, except for cured cervical carcinoma in situ, ductal carcinoma in situ of the breast, prostatic intraepithelial neoplasia, superficial non-invasive bladder cancer, stage I skin cancer (except melanoma); subjects without recurrence or metastasis for > 3 years after treatment, without current evidence of tumor, and without significant risk of recurrence of previous malignant diseases in the opinion of the study doctor may also be enrolled;
* Serious allergy to the investigational drug or excipients (such as microcrystalline cellulose, etc.);
* Patients with previous (≤ 6 months before the initiation of treatment) or current severe autoimmune diseases (including adverse reactions caused by previous anti- tumor immunotherapies), or autoimmune diseases requiring long-term systemic hormone therapy at immunosuppressive dose levels (prednisone > 10 mg/day or equivalent drugs);
* HIV, hepatitis B virus(HBV), or hepatitis C virus(HCV) positive;
* Previous (≤ 6 months prior to the first dose) or current evidence of the following diseases: acute myocardial infarction, unstable angina and cerebrovascular accident;
* Subjects who have impaired cardiac functions or clinically significant cardiac diseases;
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
recommended phase-2 dose (RP2D). | Approximately 2 years
  RP2D should be selected based on a comprehensive assessment of maximum tolerated dose(MTD), toxicity, pharmacokinetic(PK) profile, and efficacy data.
Number of participants with dose limiting toxicities | Approximately 2 years
  Dose-limiting toxicity (DLT) is defined as an adverse event (AE) or clinically significant abnormal laboratory value occurring in Cycle 1 (DLT assessment period), which is unrelated to progressive disease, concurrent disease, or concomitant medication but related to JAB-21822 and/or JAB-3312, and meets the criteria for DLT.

SECONDARY OUTCOMES:
Number of participants with AEs | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of AEs and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imagings and ophthalmological assessments
Objective response rate (ORR) | Approximately 2 years
  ORR is defined as the proportion of participants with confirmed complete response or partial response
Progression-free survival (PFS) | Approximately 2 years
  Period of time from the start of treatment to tumor progression or death from any cause (whichever occurs first) based on RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Wang Wang Jie M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (27):
- China (27):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - Pecking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy Of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Captal Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Xiamen University, Xiamen, Fujian
  - The first Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southem Medical University, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy Of medical Sciences Shenzhen Center, Shenzhen, Guangdong
  - Harbin Medical University Cancer Hospital-Mammary gland of internal, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hosipital Of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital Central South Univesity, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - The Affilated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Zhejiang School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhong J, Zhao J, Duan J, Fang J, Fei K, Li X, Chen J, Wang Z, Chu Q, Yu Y, Liu Z, Zhang L, Zhao Y, Li X, Wu L, Xing L, Zhuang W, Fang X, Chang J, Pan Y, Dong X, Liu L, Bai C, Pan P, Song Q, Jin B, Cao B, Ye F, Shi J, Tang K, Wang-Gillam A, Ding Y, Bi C, Shao Y, Pang J, Wan R, Sun B, Xu J, Wang J; JAB-21822-1006 Study Group. Glecirasib plus sitneprotafib in patients with KRASG12C-mutated non-small-cell lung cancer in China: an open-label, multicentre, single-arm, phase 1/2a trial. Lancet Respir Med. 2025 Nov 28:S2213-2600(25)00258-9. doi: 10.1016/S2213-2600(25)00258-9. Online ahead of print. PMID 41325755
- [Derived] Kang D, Wang Y, Lin Y, Ma WW, Morgensztern D, Leventakos K, Bi C, Ding Y, Xiong J, Yan M, Sun X, Wang P, Ma C, Wang Y. JAB-3312, a Potent Allosteric SHP2 Inhibitor That Enhances the Efficacy of RTK/RAS/MAPK and PD-1 Blockade Therapies. Clin Cancer Res. 2025 Jul 15;31(14):3019-3032. doi: 10.1158/1078-0432.CCR-24-3691. PMID 40333694